CLINICAL TRIAL: NCT01630096
Title: COLITIS: Clostridial Infection and Oral Lavage -Improving Treatment Before Illness Becomes Severe
Brief Title: Clostridial Infection and Oral Lavage -Improving Treatment Before Illness Becomes Severe
Acronym: COLITIS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ascension Health (Industry)
Responsible Party: Principal Investigator, Mark Vance, DO, Attending Surgeon, Ascension Health
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: GRMC 12 0008
Record Dates: First submitted 2012-06-21; First posted 2012-06-28 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Clostridium Difficile Colitis
MeSH Terms: conditions — Enterocolitis, Pseudomembranous | interventions — polyethylene glycol 3350

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nu-Lytely (Active Comparator): Bowel prep solution.
  Interventions: Drug: Nu-Lytely
- Control (No Intervention): Standard of care.

INTERVENTIONS:
Drug: Nu-Lytely — Bowl prep solution.
  Other Names: Polyethylene Glycol 3350; PEG 3350
  Arms: Nu-Lytely

SUMMARY:
Once the lab test is positive for c. diff, the investigators will order the patient to have PEG 3350 solution, one 8oz glass every ten minutes until 6 liters are gone, but if still not clear 2 more liters may be ordered. At enrollment, the treatment arm will have an order for 500 cc Normal saline to be given I.V. The patient will continue with antibiotic treatment as well. The investigators will plan to check c. diff tests daily to see when they become negative. The investigators will perform chart audit/review to track mortality, the length of stay, ICU days, surgical intervention, and APACHE scores (assessment of disease severity). Chart audit will be used to collect data on their diet and how they feel using a visual analog scale (collected by nursing staff daily as a standard procedure; see attached pain scale). Using chart audit, the investigators will record whether the patient is immunocompromised or not.

DETAILED DESCRIPTION:
Project Summary:

Clostridium Difficile (c. diff) is a bacteria which causes much morbidity and mortality worldwide. It does so by causing diarrhea and abdominal pain. It can be mild and self-limited, to severe and lethal, even in developed countries. It can require removal of the colon to try to spare a victim's life. This isn't always successful. Current treatment is withdrawal of any unnecessary antibiotics, addition of one of two antibiotics that work pretty reliably against c.diff, hydration, and observation for signs the patient might need to be operated.

The investigators propose that instead of trying to kill the bacteria that are a problem, with limited antibiotic choices, the investigators can give the patient a bowel prep and quickly and reliably wash the bacteria, and the toxin that actually wreaks the havoc, out of their system.

The investigators will collect variables of mortality, LOS, ICU days, surgical interventions (colectomy or ileostomy and lavage), time to test negative after treatment starts, and APACHE scores. The investigators will track when regular diet is resumed. The investigators will track immunocompromised state and see the effect it has. The investigators will use a visual analog scale to assess time to feel better as well.

Project description:

Rationale- Clostridium difficile (c. diff) is a bacteria in the gut which has the ability to make us very sick by releasing toxins which cause colitis. It has traditionally affected the hospitalized and those who have recently had antibiotics. Recently the investigators have seen more community acquired cases as well as cases with no antibiotics preceding the infection. C. diff can produce self-limited diarrhea and bloating, or become very severe and include severe diarrhea, bowel necrosis, toxemia and death. Over the last four years at Genesys, death rates with c. diff (all cause mortality rates) have averaged 9.6% of those infected. The investigators have averaged over 230 cases per year of c. diff infections. Clearly this is a big problem.

Traditional treatment is IV fluids, one of two antibiotics (vancomycin or flagyl) along with bowel rest, and withdrawing any unnecessary broad spectrum antibiotics (Cohen, 2010.) This helps most people, but can still progress in some cases. If the disease is or becomes severe enough, near total colon resection is required (surgery), but by that point in the disease process, 35-80% will die anyway (Neal, 2011.) Those that survive have a lot of morbidity from the ileostomy they now have (the hassle of stooling into a bag, and the dehydration that frequently accompanies the ileostomy). It's an extremely challenging problem which should be feared to worsen if and when it becomes resistant to the very few antibiotics that are currently effective. The investigators need to find a better way to treat it.

Recently out of Pittsburgh, a study was performed in which they took very sick patients to the operating room earlier and diverted the stool stream with an ileostomy and flushed Go-Lytely (polyethylene glycol) through the colon to clean it out of all the stool, bacteria, and toxin (but did not remove the colon), followed by antibiotics through the colon. They showed a reduction in the mortality rate after surgery from 50% down to 19% for a reduction of 62% (Neal, 2011). The results are very promising, but this process does require two operations - one to make the ileostomy and another to reverse the ileostomy later on. It also waits until the patients get very sick to clean out the GI tract of the bacteria and toxin.

A second paper reported two cases of chronic c. diff patients taking a bowel prep of Go-Lytely by mouth, and then being 'cured' after 36-48 months and counting (Liacouras, 1996).

In the investigators study, the investigators will still withdraw any unnecessary antibiotics, provide hydration, and treat with the same antibiotic regimen the admitting physician has decided on. But the investigators will also add a bowel prep of polyethylene glycol 3350 solution (PEG solution), to flush out the stool and bacteria. The investigators suspicion is that by giving c. diff patients a bowel prep of PEG solution orally (or nasogastric tube if unable to swallow), the investigators can wash out the c. diff bacteria and toxin they have already produced, instead of trying to kill the bacteria still in the colon. The investigators think the investigators can effectively treat even sick c. diff patients without an operation. In fact, the investigators can quite possibly prevent many mild cases from progressing to severe cases in the first place, thereby greatly decreasing the morbidity and mortality of this scary disease.

Objective- The investigators primary objective is to show that oral administration of polyethylene glycol bowel prep solution decreases mortality in clostridium difficile infected patients. Secondary objectives include showing decreased length of hospital stay, decreased ICU days, decreased time to test negative for c. diff toxin in the stool, and decreased surgical interventions, and better patient perceptions. The investigators will use a visual analog scale to track how quickly patients perceive they are better. The investigators will also determine if timing of diet resumption or immunocompromised status changes outcomes in the study.

Methodology- The study will be a prospective, randomized, controlled trial. Eligible patients will be assigned by a computer generated, randomized list to either standard treatment (IV fluids and vancomycin or flagyl) or the intervention treatment (IV fluids, vancomycin or flagyl, and oral bowel prep).

Study subject criteria includes: all adults greater than age 18, testing positive for c. diff as GRMC inpatients. Testing will be via either DNA amplification assay, or through flexible endoscopic diagnosis. The lab or endoscopist will contact Dr. Vance or Dr. Alvarez, and they will approach the patient to then consent, enroll, and randomize them.

There are no sex or ethnic background exclusion criteria, and health status of the patient will not alter patient selection. The investigators plan to enroll a total of 400 subjects.

Exclusion criteria include:

1. Pregnancy
2. Less than 18 yrs of age
3. Mentally handicapped
4. Those sick enough to require surgery at diagnosis shall not be enrolled, as they should be operated at that point.
5. Patients in whom severe ileus or suspected small bowel obstruction is present.

Interventions- Nu-Lytely or Go-Lytely (polyethylene glycol 3350), produced by Braintree Laboratories, Incorporated, will be administered to the study patients. These two products are interchangeable at the investigators institution and work by the same mechanism of action as a mechanical bowel prep. They will be dosed at one 8oz glass, orally, every 10 minutes until 6 liters are ingested. If they are not having clear bowel movements at that point, then 2 more liters will be given. If there is difficulty drinking the solution, the investigators will offer to place a nasogastric tube to deliver the PEG solution to the GI tract. It is FDA approved for bowel cleansing, though not specifically for clearing c.diff. It has a long history of effective bowel prepping with good patient safety.

Because the PEG solution can be dehydrating to a degree, the investigators will plan to give a 500 mL IV bolus of saline with the start of the bowel prep to prevent this from being an issue. These patients are generally dehydrated from the disease process anyway, and IV fluids are generally a good idea. The investigators will monitor the patients' BUN and creatinine, blood pressure, heart rate, and urine output and treat additionally for dehydration as needed.

If a patient's electrolytes are significantly abnormal at enrollment, the investigators may order an additional chemistry panel that evening to ensure this is not worsening. The investigators expect this would already be ordered by the primary physician in most cases, even without the PEG solution, in routine patient care.

To accomplish the investigators secondary objective of time to test negative for c. diff, the investigators will also collect stool to test for c. diff daily, starting the day after enrollment until negative. This will be the Immuno card c. diff toxins A& B test (available from Meridian Bioscience), as the DNA amplification method can yield false positive results with bowel preps.

Observations- The observations made by chart review after discharge will include mortality, length of stay, operative interventions, and presenting APACHE scores. Time to test negative after treatment starts will be assessed daily, and be based on stool testing results. Diet will be at the admitting physicians' discretion based on the patient status, but the investigators will monitor to see if it seems to affect successes in treating the c. diff. Additionally, the investigators will use a visual analog scale to determine when patients feel better. Nurses are required by standing policy to record visual analog pain scale responses (scale is attached). The investigators will use these responses for the study.

Sample size- To show that a mortality reduction of 70% is significant in a population with 10% mortality, a power analysis determined that 200 in each group is required to achieve 82% power detection. A total of 400 subjects will be enrolled into the study.

Data Management and Analysis- The primary hypothesis of comparing mortality between groups will be conducted using Chi square analysis. The secondary hypothesis of comparing mean days to negative test for c. diff toxin, will be analyzed using the Independent Students' t-Test for means (Mann Whitney-U test for comparing median number of days). Hospital and ICU LOS will be compared using Students' t-Test and patient perceived improvement will be compared using the Mann Whitney-U test. Surgical intervention rate will be compared by group with Chi-square analysis.

Ethical Considerations:

The study is ethical based on the possibility of a more effective way to treat a difficult disease, and the possibility of decreasing the patients' own mortality and rate of surgical interventions. The possible nausea, dehydration, abdominal bloating and discomfort will be treated symptomatically, and the rewards potentially much outweigh the risks.

Persons with mental disabilities will be excluded. If the study is a success, this may dramatically reduce mortality at Genesys and elsewhere. The Centers for Disease Control estimates that over 14,000 patients die in the USA annually from c.diff infection induced diarrhea. The investigators couldn't locate worldwide numbers, but clearly significant, and a reduction in those deaths through an effective, widely available, inexpensive treatment should be welcome everywhere.

Informed decision-making:

Study eligible patients will be approached by the study physicians. The study will be explained to the patient and their family when present. The consent form will be provided to the patient and they will be given time to ask questions and read over the consent form. The investigators informed consent form is attached. Patients who agree will be enrolled into the study by the study physicians.

Gender Issues:

The investigators plan to include women and men alike in the study. When the investigators analyze the data, the investigators will determine any significant differences in outcomes based on gender, and report these.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older male or female testing positive for c. diff

Exclusion Criteria:

* Pregnancy Less than 18 yrs of age Those sick enough to require surgery at diagnosis Severe ileus or small bowel obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Length of stay | 30 days
  Days

SECONDARY OUTCOMES:
Need for surgery | 30 days
  Did the subject have an operation, if so what was it (colectomy/illeostomy&lavage).

CONTACTS AND LOCATIONS:
Overall Officials: Mark B. Vance, DO, Principal Investigator — GRMC
Locations (1):
- Genesys Regional Medical Center, Grand Blanc, Michigan, United States